CLINICAL TRIAL: NCT04796493
Title: Is Objective Grading of Mesenteric Traction Syndrome With Laser Speckle Contrast Imaging Interchangeable With Digital Thermography
Brief Title: Objective Grading of MTS With LSCI and Thermography
Acronym: MTS LSCI
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, August Adelsten Olsen, MD PhD student, Rigshospitalet, Denmark
Other Study IDs: H-20058773
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Mesenteric Traction Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Mesenteric traction syndrome (MTS) is defined as hypotension, tachycardia and facial flushing in the first hour of surgery, caused by mesenteric traction/abdominal exploration. MTS occurs frequently during abdominal surgery, with incidence around 80 % during open surgery, and lower during minimally invasive surgery. MTS can be divided into different severities using the degree of facial flushing, with the most severe level of MTS being associated with increased postoperative morbidity.

Today MTS is diagnosed and graded subjectively by the surgical team, with marked difficulty and limitations. Therefore the investigators developed a cut-off value using the Laser Speckle Contrast Imaging (LSCI), which the investigators wish to confirm in a new cohort, while also examining whether LSCI is interchangeable with digital thermography, which is simpler and cheaper to perfom.

The investigators will measure facial perfusion during the first hour of surgery and take blood samples at predefined timepoints to use for biochemical verification of the different severities of MTS.

Three cohorts we planned to include 45 open esophagectomies or gastrectomies 50 whipple surgery 20 robot assisted esophagectomies or gastrectomies These patients will be use in multiple articles examining different aspects of MTS

One study examining LSCI and thermography for the identification and grading of MTS will use 60 patients undergoing open esophagectomy or gastrectomy or whipple surgery, in this study patients will not be excluded if they are found to be disseminated.

However we ended up including 37 open esophagectomies - due to few patients undergoing open esophagectomy, this were included over a time period of almost 2,5 years 50 whipple 11 Robotic esophagectomies - due to LSCI being impossible to use on robotic esophagectomies and thermography being diffciult to fit on these patients and as such not being feasible

ELIGIBILITY:
Inclusion Criteria:

* Undergoing curative surgery for esopageal, gastric, doudenal or pancreatic cancer

Exclusion Criteria:

* Known flushing disease
* Patients recieving NSAID and corticosteroid presurgery, Whipple is allowed to recieve single dose of 125 mg Methylprednisone as part of the standard of care at our facility.
* Palliative surgery
* Surgery not completed due to disseminated disease - patients will still be used in examination of LSCI and Thermography analysis even if desiminated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3 cohorts
  * open esophagectomies
  * robotic assisted esophagectomies
  * whipples procedure
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2027-08-23 (Estimated)

PRIMARY OUTCOMES:
Severity of MTS - measured facial perfusion | first hour of surgery
  Facial perfusion measured with LSCI and Digital Thermography

SECONDARY OUTCOMES:
Biochemical markers of MTS - prostacyclin | During surgery
Hemodynamics | During surgery
Markers of postoperative impact of MTS - IL6 and endothelial damage markers | During and after surgery
30-day postoperative morbidity | 30 days post surgery
Incidence of objective MTS during whipples procedure with methylprednisolone prophylaxis | During surgery
Incidence of objective MTS during minimally invasive surgery | during surgery
PACU - fluid therapy administred at PACU | At the PostAnesthesia Care Unit following surgery. Typically one to two days
PACU - vasopressor requirements | At the PostAnesthesia Care Unit following surgery.Typically one to two days
PACU - length of stay | At the PostAnesthesia Care Unit following surgery. Typically one to two days
suPAR (soluble urokinase Plasminogen Activator Receptor). | baseline just prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: August Olsen, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, København Ø, Capital Region, Denmark